CLINICAL TRIAL: NCT04349878
Title: Effect of Phytotherapy Agens in Non Surgical Periodontitis
Brief Title: Anaysis of Phytotherapy Agent Against Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Assistant professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-2018
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): scaling and root planing alone
  Interventions: Diagnostic Test: gingival crevicular fluid evaluation
- phytotherapeutic (Active Comparator): scaling and root planing plus phytotherapeutic agent
  Interventions: Diagnostic Test: gingival crevicular fluid evaluation

INTERVENTIONS:
Diagnostic Test: gingival crevicular fluid evaluation — anaysis of interleukins in gingival crevicular fluid

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence of the decontaminant tools for the management of Periodontitis (, the aim of this study was to evaluate, at 6 months follow-up, the post-treatment clinical parameters and immunological and gingival microbial profiles in patients with periodontitis, treated by either SRP in addition to phytotherapeutic drug or SRP alone.

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2008. The local ethical committee of the University of Messina approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent 34 patients, 18 men and 16 women, aged 27 to 65 (mean age 44.2) were assessed for eligibility . In all subjects, subgingival plaque was acquired from 4 separate proximal sites at 365 days after therapy.

The Gingival Crevicular Fluid (GCF) was gathered, at the same time from other four different non-contiguous interproximal sites using filter paper strips‡ as previously described. The levels of IL-1β, IL-10 and TNF-α were recognized by conventional enzyme-linked immunosorbent assay using an equation with software using a five polynomial parameter. Each selected subject underwent randomly, without anaesthesia, at the same time and after recording periodontal parameters, the two following treatments: in one, were treated as conventional Scaling and Root Planing (SRP) + phytotherapeutic drug (Neuridase), while the other group were treated as conventional SRP alone

ELIGIBILITY:
Inclusion Criteria:

1. good condition of general health,
2. a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm,
3. no involvement of the furcation,
4. a minimum of a six teeth per quadrant, respectively.

Exclusion Criteria:

1. periodontal therapy during the last 12 months,
2. assumption of antibiotics during the last 6 months,
3. pregnancy,
4. any systemic condition which might affect the effects of the study treatment,
5. previous or current radiation or immunosuppressive therapies,
6. use of mouthwash containing antimicrobials during the previous 3 months,
7. no use of hormonal contraceptives,
8. medication by anti-inflammatory and immunosuppressive drugs,
9. previous history of hard-drinking,
10. smoking,
11. class II and III tooth mobility.

Ages: 32 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment level | 180 days
  Analysis of reduction of clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Gatano Isola, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing inflammatory results
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: University website and pubmed